CLINICAL TRIAL: NCT00884104
Title: A Prospective, Open-label, Observational, Multi-center Study for the Identification of Predictive Factors for the Solifenacin Treatment in Men With Overactive Bladder Symptoms After Tamsulosin Monotherapy for 4 Weeks and Evaluation of Efficacy and Persistency of Add on Solifenacin in Men With Residual Overactive Bladder Symptoms After Previous Monotherapy With Tamsulosin.
Brief Title: A Study to Evaluate Add on Effect of Solifenacin in Men With Overactive Bladder Symptoms After Tamsulosin Monotherapy for 4 Weeks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KYU-SUNG LEE (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor-Investigator, KYU-SUNG LEE, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMK-3
Record Dates: First submitted 2009-03-25; First posted 2009-04-20 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Overactive Bladder
Keywords: Solifenacin; Tamsulosin; OAB
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1.tamsulosin + solifenacin (Experimental)
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Solifenacin — Oral
  Other Names: Vesicare

SUMMARY:
The purpose of this study is to evaluate the rate of "add-on" solifenacin treatment and its persistency in men with over active bladder symptoms after tamsulosin monotherapy for 4 weeks.

DETAILED DESCRIPTION:
This is a multi-center study to evaluate the efficacy, safety, and persistency of solifenacin treatment in male patients with persistent OAB symptoms of urinary frequency and urgency with/without urgency incontinence who are receiving tamsulosin monotherapy for LUTS at a stable dose for 4 weeks in real life practice. Also proportion of patients and predictive factors with persistent OAB symptoms after tamsulosin monotherapy will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* IPSS ≥ 12
* Symptoms of OAB as verified by the V8 (≥8)
* Symptoms of OAB as verified by the screening 3-day bladder diary, defined by:

  * Mean urinary frequency ≥8 times/24 hours
  * Mean number of micturition-related urgency episodes ≥3 episode/24 hours (with a Urinary Sensation Scale rating of ≥3 marked for the corresponding micturition in the bladder diary)

Exclusion Criteria:

* Treatment within the 14 days preceding treatment with any alpha blocker drugs
* A known history of bladder outlet obstruction due to: bladder neck contracture, clinical suspicion of prostate carcinoma, mullerian duct cysts, urethral obstruction due to stricture/valves/sclerosis or urethral tumor

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with "add-on" solifenacin treatment | Weeks of 12, 24 and 52 of combination therapy

SECONDARY OUTCOMES:
Change from baseline in micturition efficacy parameters | Weeks of 12, 24 and 52 of combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, MD, Principal Investigator — University School of Medicine, Kangnan-ku, Seoul, Korea
Locations (9):
- South Korea (9):
  - Cheonju
  - Choongju
  - Daegu
  - Daejeon
  - Kangneung
  - Kwangju
  - Pusan
  - Seoul
  - Suwon

REFERENCES:
- [Derived] Lee HN, Lee KS, Kim JC, Chung BH, Kim CS, Lee JG, Kim DK, Park CH, Park JK, Hong SJ. Rate and associated factors of solifenacin add-on after tamsulosin monotherapy in men with voiding and storage lower urinary tract symptoms. Int J Clin Pract. 2015 Apr;69(4):444-53. doi: 10.1111/ijcp.12581. Epub 2014 Nov 1. PMID 25363606